CLINICAL TRIAL: NCT04752631
Title: MRI-guided thrOmbolysis for Stroke bEyond Time Window by TNK (ROSE-TNK): a Prospective, Randomized, Blinded Assessment of Outcome and Open Label Multi-center Study
Brief Title: MRI-guided thrOmbolysis for Stroke bEyond Time Window by TNK
Acronym: ROSE-TNK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of neurology department, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y(2020)067
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Stroke
Keywords: TNK-tPA; stroke
MeSH Terms: conditions — Stroke | interventions — Tenecteplase; TNK-tissue plasminogen activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Outcomes will be performed by a blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNK-tPA (Experimental): TNK-tPA (0.25mg/kg) given as a single bolus over 5-10 seconds immediately upon randomization.
  Interventions: Drug: Tenecteplase
- Routine Therapy (No Intervention): Patients will be treated with standard of care in compliance with guidelines for acute stroke

INTERVENTIONS:
Drug: Tenecteplase — The participants received TNK-tPA thrombolytic therapy
  Other Names: TNK-tPA
  Arms: TNK-tPA

SUMMARY:
This is an open label multicentre trial, evaluating the utility of MRI-guided thrombolysis for stroke beyond time window by Tenecteplase (TNK-tPA). This exploratory study was to describe the feasibility and outcome of thrombolytic therapy with TNK-tPA in 4.5-24 hours after stroke guided by a mismatch between diffusion-weighted imaging and FLAIR in the region of ischemia.

DETAILED DESCRIPTION:
In patients with acute stroke with an unknown time of onset, intravenous alteplase guided by a mismatch between diffusion-weighted imaging and FLAIR in the region of ischemia resulted in a significantly better functional outcome at 90 days. This trial will enroll acute ischemic stroke patients within 4.5 to 24 hours of onset. All the patients had an ischemic lesion that was visible on MRI diffusion-weighted imaging but no parenchymal hyperintensity on fluid-attenuated inversion recovery (FLAIR), which indicated that the stroke had a ischemic penumbra. Randomization will be 1:1 to TNK-tPA (experimental) or standard treatment (control), in compliance with guidelines for acute stroke. Clinical outcome was assessed by disability on the basis of the modified Rankin scale at 90 days follow-up, which will be performed by a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18-80 years;
2. The time from onset to treatment: 4.5-24 hours;
3. Acute Ischemic stroke confirmed by MRI;
4. NIHSS score ：6-25, or NIHSS score≤ 5 but culprit vessel occlusion or severe stenosis ( ICA, MCA-M1/M2, ACA) on CTA/MRA;
5. Imaging requirements: (1) DWI infarct region: no more than 1/3 of middle cerebral artery territory or 1/2 of the anterior cerebral artery territory or 1/2 of the posterior cerebral artery territory; (2) DWI infarct volume <70 ml; (2) presence of DWI/Flair mismatch: DWI high signal and Flair visually normal;
6. the first onset of ischemic stroke or previous stroke with no obvious sequelae (mRS≤1);
7. Signed informed consent

Exclusion Criteria:

1. Planned endovascular treatment;
2. Serious neurological deficits before onset ( mRS ≥ 2);
3. Obvious head injuries or strokes within 3 months;
4. Subarachnoid hemorrhage;
5. History of intracranial hemorrhage;
6. Intracranial tumor, arteriovenous malformation or aneurysm;
7. Intracranial or spinal cord surgery within 3 months;
8. Arterial puncture at a noncompressible site within the previous seven days;
9. Active internal hemorrhage;
10. coagulation abnormalities: platelet count of <100000/mm3 ；
11. Aortic arch dissection；
12. Heparin therapy within 24 hours;
13. Infective endocarditis；
14. Oral warfarin is being taken and INR>1.6 or APTT abnormal；
15. oral anticoagulation therapy；
16. Systolic pressure ≥185 mmHg or diastolic pressure ≥110 mmHg；
17. Blood glucose < 50 mg/dl (2.7mmol/L)；
18. Pregnancy;
19. Neurological deficit after epileptic seizures;
20. Major surgery within 1 month;
21. Gastrointestinal or urinary tract hemorrhage within the previous 30 days;
22. Myocardial infarction within 3 months;
23. allergy to study drugs;
24. Contradictory to MRI examination；
25. MRI image not qualified for evaluation；
26. Other serious illness；
27. Participating in other clinical trials within 3 months;
28. patients not suitable for this clinical studies considered by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
Proportion of modified Rankin Scale (mRS) 0-1 | 90 Days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome

SECONDARY OUTCOMES:
Proportion of modified Rankin Scale (mRS) 0-2 | 90 Days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome
Distribution of the modified Rankin Scale (mRS) | 90 Days
  the minimum and maximum values of mRS are 0 and 6, respectively; higher mRS mean a worse outcome
Changes in National Institute of Health stroke scale (NIHSS) | 24 hours and 1 week
  the minimum and maximum values of NIHSS are 42 and 0, respectively; higher NIHSS mean a worse outcome
vascular events | 90 Days
  The incidence of stroke and other vascular events
proportion of death | 14 days
  death due to any cause

OTHER OUTCOMES:
Proportion of symptomatic intracranial hemorrhage (sICH) | 48 hours
  sICH was defined as 4 or more increase in NIHSS caused by hemorrhage
Proportion of intraparenchymal hemorrhage (PH1 and PH2) | 48 hours
  Proportion of PH1 and PH2 within 48 hours after the treatment
proportion of hemorrhagic transformation | 7 Days
  Intracranial hemorrhage assessed by MRI/CT
any bleeding events | 7 Days
  proportion of any bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Chen Hui-Sheng, Doctor, Study Director — General Hospital of Shenyang Military Region
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomalla G, Simonsen CZ, Boutitie F, Andersen G, Berthezene Y, Cheng B, Cheripelli B, Cho TH, Fazekas F, Fiehler J, Ford I, Galinovic I, Gellissen S, Golsari A, Gregori J, Gunther M, Guibernau J, Hausler KG, Hennerici M, Kemmling A, Marstrand J, Modrau B, Neeb L, Perez de la Ossa N, Puig J, Ringleb P, Roy P, Scheel E, Schonewille W, Serena J, Sunaert S, Villringer K, Wouters A, Thijs V, Ebinger M, Endres M, Fiebach JB, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Gerloff C; WAKE-UP Investigators. MRI-Guided Thrombolysis for Stroke with Unknown Time of Onset. N Engl J Med. 2018 Aug 16;379(7):611-622. doi: 10.1056/NEJMoa1804355. Epub 2018 May 16. PMID 29766770